CLINICAL TRIAL: NCT01362998
Title: A Comparison of Single Dose Preservative Free Morphine With Fentanyl Infusion for Post-Cesarean Section Analgesia
Brief Title: Epidural Morphine Versus Epidural Fentanyl Infusion Following Cesarean Section
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of time and help to continue the study
Sponsor: Goodman, Evan, M.D. (Individual)
Responsible Party: Principal Investigator, Dr. Evan Goodman, MD, Anesthesiologist, Goodman, Evan, M.D.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: goodman-2
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Pain
Keywords: fentanyl, morphine, duramorph, Cesarean section, epidural
MeSH Terms: conditions — Pain | interventions — Morphine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preservative free morphine (Active Comparator): This group will receive 3mg of preservative free morphine epidurally during the procedure.
  Interventions: Drug: Preservative free morphine
- Fentanyl infusion (Active Comparator): This group will receive an epidural infusion of fentanyl (60 micrograms per hour), which will be started during the Cesarean section and which will continue for the next two days.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Preservative free morphine — 3mg given epidurally during the Cesarean section.
  Other Names: Duramorph
  Arms: Preservative free morphine
Drug: Fentanyl — An infusion of epidural fentanyl started during the Cesarean section. It will be given on a patient controlled analgesia basis, with a basal rate of 60 micrograms, a demand dose of 16 micrograms, and a lockout of 15 mins.
  Other Names: PCA fentanyl
  Arms: Fentanyl infusion

SUMMARY:
For post-Cesarean analgesia, the investigators will compare the efficacy of single-shot epidural preservative free morphine with a continuous epidural fentanyl infusion. The investigators will be comparing the patient's pain level and satisfaction with the two techniques, as well as the side effects that the patients experience, such as itching, nausea, back pain and respiratory depression.

DETAILED DESCRIPTION:
Included in the study will be all healthy (ASA I or II) woman having elective Cesarean sections who are candidates for regional anesthesia. Exclusion criteria include morbid obesity (BMI > 40), age less that 18 years, history of sleep apnea, and abuse of or intolerance to opioid analgesics.

All patients will also receive 100 micrograms of fentanyl once epidurally during the Cesarean section, and they will receive ibuprofen every six hours for the first 24 hours after the Cesarean section. The patients will be visited twice a day postoperatively for two days. The epidural morphine will be expected to last only approximately 20 hours, while the fentanyl infusion will be kept in place for two days after the procedure. Additional analgesics, such as intravenous morphine or PO oxycodone and tylenol, will be available for breakthrough pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients having an elective Cesarean section
* Healthy women (ASA I or II)
* Regional anesthesia candidates

Exclusion Criteria:

* Morbid obesity (BMI>40)
* Sleep apnea
* Age under 18
* Intolerance or addiction to opioids

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Goodman, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Sarvela J, Halonen P, Soikkeli A, Korttila K. A double-blinded, randomized comparison of intrathecal and epidural morphine for elective cesarean delivery. Anesth Analg. 2002 Aug;95(2):436-40, table of contents. doi: 10.1097/00000539-200208000-00037. PMID 12145067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 people were recruited for this study, but data was collected for only one of them.
Period: Overall Study
Arm/Group | Preservative Free Morphine | Fentanyl Infusion
Started | 0 | 2
Completed | 0 (Note: No participants in this arm.) | 1
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Note that no people were recruited for the morphine arm. Note that 2 people were recruited for the fentanyl arm, but that data was collected for only 1 person.
Groups:
- Total: Total of all reporting groups
Arm/Group | Preservative Free Morphine | Fentanyl Infusion | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: Years] |  | 27 [27 to 27] | 27 [27 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Weight, continuous [Number; unit: pounds] |  | 179 | 179
Pregnancies, integer [Number; unit: Number of pregnancies] |  | 4 | 4
Gestational age, continuous [Number; unit: Weeks] |  | 39 | 39

OUTCOME MEASURES:

1. Primary Outcome: Postsurgical Pain
Description: Participants will be asked to rate their pain on a 10 point Numerical Rating Pain Scale, where zero is no pain and ten is the most intense pain possible.
Time Frame: At 8, 24 36 and 48 hours after the Cesarean section
Population: No participants in morphine arm.
Measure: Number; unit: Units on a 10 point scale
Arm/Group | Preservative Free Morphine | Fentanyl Infusion
Number analyzed (Participants) | 0 | 1
Units on a 10 point scale
  8 hours post Cesarean section |  | 3
  24 hours post Cesarean |  | 0
  36 hours post Cesarean |  | 3
  48 hours post Cesarean |  | 7

2. Secondary Outcome: Number of Participants Who Responded Yes to Having Nausea or Vomiting
Description: The patient will be asked whether she has nausea or vomiting (yes=1, no=0).
Time Frame: At 8, 24, 36 and 48 hours after the Cesarean section
Population: No patients were in the morphine group
Measure: Count of Participants; unit: Participants
Arm/Group | Preservative Free Morphine | Fentanyl Infusion
Number analyzed (Participants) | 0 | 1
Participants
  8 hours after the surgery |  | 0
  24 hours after the surgery |  | 0
  36 hours after the surgery |  | 0
  48 hours after the surgery |  | 0

3. Secondary Outcome: Patient Satisfaction
Description: Participants will be asked to rate their satisfaction on a 10 point Numerical Rating Scale (0=worst, 10=best).
Time Frame: At 8, 24, 48 and 36 hours after Cesarean section
Population: There were no participants in the morphine arm.
Measure: Number; unit: score on a scale
Arm/Group | Preservative Free Morphine | Fentanyl Infusion
Number analyzed (Participants) | 0 | 1
score on a scale
  8 hours after the surgery |  | 10
  24 hours after the surgery |  | 10
  36 hours after the surgery |  | 10
  48 hours after the surgery |  | 10

4. Secondary Outcome: Number of Participants Who Responded Yes to Having Back Pain
Description: Participants will be asked whether they have back pain (Yes=1, No=0)
Time Frame: At 8, 24, 36 and 48 hours after the Cesarean section
Population: No participants in the morphine arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Preservative Free Morphine | Fentanyl Infusion
Number analyzed (Participants) | 0 | 1
Participants
  8 hours after the surgery |  | 0
  24 hours after the surgery |  | 0
  36 hours after the surgery |  | 0
  48 hours after the surgery |  | 0

5. Secondary Outcome: Number of Participants Who Responded Yes to Having Pruritis
Description: Participants will be asked whether they have pruritis (Yes=1, No=0)
Time Frame: At 8, 24, 36 and 48 hours after Cesarean section
Population: No participants in the morphine arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Preservative Free Morphine | Fentanyl Infusion
Number analyzed (Participants) | 0 | 1
Participants
  8 hours after the surgery |  | 1
  24 hours after the surgery |  | 1
  36 hours after the surgery |  | 1
  48 hours after the surgery |  | 1

6. Secondary Outcome: Number of Participants Who Were Observed by Their Nurse to Have Urinary Retention
Description: Participant's nurse will be asked whether >400ml was obtained by straight cath (Y=1, No=0)
Time Frame: At 8, 24, 36 and 48 hours after Cesarean section
Population: No participants in morphine arm
Measure: Count of Participants; unit: Participants
Arm/Group | Preservative Free Morphine | Fentanyl Infusion
Number analyzed (Participants) | 0 | 1
Participants
  8 hours after the surgery |  | 0
  24 hours after the surgery |  | 0
  36 hours after the surgery |  | 0
  48 hours after the surgery |  | 0

7. Secondary Outcome: Number of Participants Who Were Observed by Their Nurse to Have Respiratory Depression
Description: Participant's chart will be examined to determine whether the respiratory rate was <8 per minute (Yes=1, No=0)
Time Frame: At 8, 24, 36 and 48 hours after the Cesarean section
Population: No participants in morphine arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Preservative Free Morphine | Fentanyl Infusion
Number analyzed (Participants) | 0 | 1
Participants
  8 hours after the surgery |  | 0
  24 hours after the surgery |  | 0
  36 hours after the surgery |  | 0
  48 hours after the surgery |  | 0

8. Other Pre Specified Outcome: Number of Participants Who Required Additional Pain Medications
Description: Participant's nurse will be asked whether the patient required additional pain medications (Yes=1, No=0)
Time Frame: At 8, 24, 36 and 48 hours after the Cesarean section
Population: No participants in morphine arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Preservative Free Morphine | Fentanyl Infusion
Number analyzed (Participants) | 0 | 1
Participants
  8 hours after the surgery |  | 0
  24 hours after the surgery |  | 0
  36 hours after the surgery |  | 0
  48 hours after the surgery |  | 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: Note that morphine arm has no participants.
Arm/Group | Preservative Free Morphine | Fentanyl Infusion
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Note that data was collected from only one participant in a two-armed study, so no statistical comparisons could be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes